CLINICAL TRIAL: NCT06902753
Title: Adaptation and Normalization of a Verbal Episodic Memory Test (16-item Free and Cued Recall / RL-RI 16) in French Sign Language
Brief Title: Adaptation and Normalization of a Verbal Episodic Memory Test in French Sign Language
Acronym: RL-RI-LSF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-A02627-40
Record Dates: First submitted 2024-12-30; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Neuropsychological Tests; Memory; Alzheimer Disease; Deafness; Sign Language; Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Deafness; Sign Language; Cognitive Dysfunction | interventions — Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healthy Deaf Signing Group (Experimental)
  Interventions: Other: Questionnaire and Physical Exam

INTERVENTIONS:
Other: Questionnaire and Physical Exam — Neuropsychological assessment:
  * Phase 1: MMS-LS (overall cognitive efficiency) + fluency tasks (verbal flexibility)
  * Phase 2: MMS-LS (if the participant did not take part in phase 1), RL-RI LSF (verbal memory), Rey Complex Figure (visuospatial abilities and visual memory), Progressive Matrices, Symbols and Code (executive functions)

SUMMARY:
To date, neuropsychological assessment of deaf signing persons is complicated by a lack of resources, especially the absence of tools available in French Sign Language (LSF). This is due to perceptual and cultural differences, and in particular the linguistic differences between French and LSF.

This lack of resources significantly hinders access to care for deaf patients, as neuropsychological assessment is often a key clinical criterion in the diagnosis of certain neurological pathologies (Alzheimer's disease in particular) and enables coherent care plans to be drawn up, for example in the aftermath of strokes or traumatic brain injuries.

In particular, episodic memory (which refers to the ability to memorise information anchored in a specific context) is a cognitive domain that is sensitive to pathologies such as Alzheimer's disease, but it is not currently possible to assess it with deaf signing patients.

The aim of this study is to create a memory assessment test adapted to a deaf population that expresses in LSF and to normalize this test on this same population.

The aim is to provide a diagnosis assessment tool, which currently does not exist in France, to improve access to care for deaf people. This project could then be extended to the creation of tests for other cognitive domains (executive functions, attention, social cognition, etc.) and to prospects for cognitive remediation.

The 16-item Free and Cued Recall test (RL-RI 16) is the best choice because it is easy to use and accurate enough to assess each stage of episodic memory. These qualities make it a decisive tool in certain differential diagnosis.

In order to select the most relevant signs, lexical lists by frequency in LSF will be drawn up during a preliminary phase, during which the participants will have to give, in one minute, the maximum number of signs belonging to different categories (animals, vegetables, clothes...). These lists will be used to select the most relevant signs according to their frequency (neither too common nor too rare), based on the same principle as RL-RI 16.

It will then be standardised on deaf adults, for whom LSF is the main language, with no cognitive impairment, across France, via the various Deaf Care Units, with the help of French / LSF interpreters. Working with different centers in France will make it possible to recruit a larger and more representative number of participants, and to be more sensitive to any regional effects.

ELIGIBILITY:
Inclusion Criteria:

* Person aged ≥ 18 yo
* with severe or profound deafness (hearing loss ≥ 70 decibels)
* whose main language is French Sign Language
* able to consent in writing after a clear explanation of the procedure
* affiliated to the French Healthcare system (Sécurité Sociale) through self or another person

Non-inclusion criteria:

* person with a medical history in neurology (stroke, traumatic brain injury, dementia) or psychiatry bipolar syndrom or schizophrenia that would not be medicated, severe depression)
* persons with medical developmental backgroung (e.g genetic syndrome)
* person with cancer history needing chemotherapy
* person with a diagnosed and untreated sleeping trouble
* person drinking > 10 glasses of alcohol per week or using drugs on a daily basis
* person with visual issues
* person under 18yo or unable to take decisions for self

Exclusion Criteria:

A score ≤ 20/28 or 17/28 at the MMS-LS test, depending on the schooling of the participant (20/28 for participants with a degree, 17/28 for participants without a degree)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Normed data for the RL-RI-LSF test for a deaf population without cognitive impairment | Phase 2: 9 months
  The main goal of this study is to propose normed data for the RL-RI-LSF test (adaptation in LSF of the RL-RI 16 test) for a deaf population without cognitive impairment.
  The RL-RI-LSF scores correspond to the number of signs correctly recalled by the patient during each recall:
  * free recalls
  * cued recalls
  * recognition scores We will model each RL-RI-LSF score as a function of the participant's gender, age and socio-cultural level. We will present an expected mean score for each age, gender and socio-cultural level class.

SECONDARY OUTCOMES:
Correlation RL-RI LSF / MMS-LS | Phase 2: 9 months
  The secondary goal is to assess the correlation of the RL-RI-LSF with the MMS-LS score
Reproductibility over time | Phase 2: 9 months
  The secondary goal is to assess the reproducibility over time (test/retest) of the RL-RI-LSF at 9-month intervals.
  The reproducibility of the RL-RI-LSF will be assessed by comparing the scores obtained at two different measurement times (RL-RI-LSF tests separated by 9 months) using the intra-class correlation coefficient.
Normative data for the Rey Complex Figure Test | Phase 2: 9 months
  The secondary goal is to propose normalised data for the Rey Complex Figure Test (visuo-spatial copying and memory test) in a French deaf-signing population without cognitive impairment.
  Each score (copy and memory, /36) will be considered and modeled, if need be, as a function of the participant's gender, age and socio-cultural level. We will present an expected mean score for each age, gender and socio-cultural level class.
Normative data for 3 subtests of the WAIS-IV | Phase 2: 9 months
  A secondary outcome is to propose normative data for 3 subtests of the WAIS-IV (Matrices, Symbols, Code) in a deaf-signing population without cognitive impairment.
  Each raw score will be considered for each test, and modeled, if need be, as a function of the participant's gender, age and socio-cultural level. We will present an expected mean score for each age, gender and socio-cultural level class.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Alexandre BERARD, Speech-Language Pathologist, Principal Investigator — Poitiers University Hospital